## Cover Page for Data Security Plan

| Sponsor Name | Northwestern University |
|---|---|
| NCT ID | NCT02357784 |
| Sponsor Trial ID | STU00098840 |
| Official Title of the study | Sacral Neuromodulation in Dual Incontinence: Ultrasound and |
| | Afferent Nerve Sensation Assessment (SaNDI) |
| Document Date | 2-8-2023 |

Each sensory modality threshold as determined at each of the different anatomic sites will be evaluated separately. Sensory thresholds will be compared before and after SNM placement using paired t-test. Multivariate regression models will be used to determine clinical and neurophysiologic predictors of symptom improvement. Urethral sphincter volumes and presence/absence and size of internal and external anal sphincter defects will be compared in responders and non-responders.